CLINICAL TRIAL: NCT06357884
Title: Short-term Effect of Podiatric Callus Debridement on Plantar Pressure in Diabetic Neuropathic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Princess Margaret Hospital, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Joanne Tze Yan LAI, MSc Student, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CREC2023.572
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Diabetic Neuropathies; Plantar Callus
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Callus debridement (Experimental): Callus debridement which aligns with routine clinical practice of the Princess Margaret Hospital Podiatry Department.
  Interventions: Procedure: Callus debridement

INTERVENTIONS:
Procedure: Callus debridement — Eligible patients will be seated on a podiatry couch. Standard skin preparation procedure will be done with 2% Chlorhexidine gluconate in 70% isopropyl cleansing to all areas of feet. The same researcher will perform sharp debridement in all participants to minimize the variance between procedures. The procedure will comply with Infection Control Guideline (Podiatry) . A sterile scalpel handle loaded with a single-use No. 15 blade will be used to carry out sharp debridement using aseptic technique. Hyperkeratotic tissue will be debrided until smooth transition with adjacent skin is achieved and underlying pinkish normal skin is visible. Used scalpel will be unloaded and disposed by a QlickSmart ® BladeFLASK scalpel blade remover.

SUMMARY:
Diabetes peripheral neuropathy (DPN) affects up to 50% of the diabetes population. In the diabetic neuropathic foot, it commonly manifests as loss of protective sensation, foot deformity and skin dryness. Alongside with day-to-day weightbearing activities, this can lead to formation of callus over plantar pressure points. Studies have proven that callus formation leads to high plantar pressure and increased risk of diabetic foot ulcers. For podiatrists, diabetic foot screening and treatment is our daily practice. Plantar callus are commonly treated by sharp debridement to relief pressure from the hard skin build up and thus reducing the risk of ulceration. However, the effectiveness of callus sharp debridement is not commonly studied in researches. Only a few studies in the past evaluated the effectiveness of callus treatment by different outcome measurements. Among those studies only 2 were specifically done in diabetic patients, in which one reported results of diabetic neuropathic patients. All the available studies used peak plantar pressure only as their pedobarographic outcome measure. In this study, the treatment effect of podiatric sharp debridement of callus in diabetic neuropathic patients will be evaluated using a range of pedobarographic parameters and Foot and Ankle Outcome Score (FAOS) questionnaire. The immediate and short-term (3-4 weeks) effect of sharp debridement in DPN patients with callus could be quantified. Change in loading pattern could also be analysed based on different areas of the foot.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Active out-patient status in Podiatry department of Princess Margaret Hospital
3. Men and women
4. Ambulatory
5. Diagnosis of type I or II diabetes
6. Failed peripheral neurological assessment (Vibration perception threshold >25 volts or unable to detect one or more sites of 4-point 10g Semmes-Weinstein monofilament test)
7. Presence of plantar callus
8. Compliance with instructions (in Chinese or english)
9. Ability to read and write (in Chinese or english)

Exclusion Criteria:

1. Peripheral vascular disease
2. Painful neuropathy
3. Charcot deformity
4. Undergone any form of callus debridement in the past 6 weeks
5. Active foot ulcer
6. Any dermatological condition other than callus that causes hyperkeratosis (e.g. verruca pedis, eczema, tinea pedis)
7. Any musculoskeletal condition that affects balance and gait
8. Allergic to chlorhexidine gluconate or alcohol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-02-23 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Peak plantar pressure (PPP) (unit: kPa) | Before treatment, immediately after treatment and 3-4 weeks post-treatment
  The maximum or highest pressure within foot

SECONDARY OUTCOMES:
Pressure time integral (PTI) (unit: kPa*sec) | Before treatment, immediately after treatment and 3-4 weeks post-treatment
  The amount of pressure relative to the time that the pressure is present
Peak pressure gradient (PPG) (unit: kPa/cm) | Before treatment, immediately after treatment and 3-4 weeks post-treatment
  Spatial change in pressure around location of the peak pressure
Forefoot to rearfoot peak pressure ratio (F/R ratio) | Before treatment, immediately after treatment and 3-4 weeks post-treatment
  Forefoot to rearfoot peak plantar pressure ratio
Foot and Ankle Outcome Score (FAOS) | Before treatment, 1 week after treatment and 3-4 weeks post-treatment
  Patient-reported outcome measurement (PROM) tool that is calculated using 42 Likert scale questions which are organised into 5 sub-categories: symptoms, pain, activities of daily living (ADL), sports and quality of life (QOL)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Ka-Kin Ling, Study Director — Assistant Professor (Clinical) of Orthopaedics & Traumatology
Locations (1):
- Podiatry Department, Princess Margaret Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No